CLINICAL TRIAL: NCT07008638
Title: HM2024-29: Phase I/II Clinical Trial of Proteasome Inhibitor in Combination With CPX-351 for the Treatment of Newly-Diagnosed TP53-mutated Acute Myeloid Leukemia (AML)
Brief Title: Phase I/II Clinical Trial of Proteasome Inhibitor in Combination With CPX-351 for the Treatment of Newly-Diagnosed TP53-mutated Acute Myeloid Leukemia (AML)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024LS157
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia; TP53
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Bortezomib; CPX-351; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1: Dose Level -1 (Experimental): Bortezomib 0.7mg/m2 in combination with CPX-351
  Interventions: Drug: Bortezomib; Drug: CPX-351
- Phase 1: Dose Level 2 (Experimental): Bortezomib 1mg/m2 in combination with CPX-351
  Interventions: Drug: Bortezomib; Drug: CPX-351
- Phase 1: Dose Level 3 (Experimental): Bortezomib 1.3 mg/m2 in combination with CPX-351
  Interventions: Drug: Bortezomib; Drug: CPX-351
- Phase 1: Dose Level 4 (Experimental): Bortezomib 1.5 mg/m2 in combination with CPX-351
  Interventions: Drug: Bortezomib; Drug: CPX-351
- Phase 2 (Experimental): Maximum tolerated dose of Bortezomib in combination with CPX-351
  Interventions: Drug: Bortezomib; Drug: CPX-351

INTERVENTIONS:
Drug: Bortezomib — Bortezomib at assigned study dose in mg/m2 will be given subcutaneously on days 1, 4, 8, and 11
Drug: CPX-351 — CPX-351 given intravenously on day 1, 3, and 5
  Other Names: Liposomal daunorubicin; Cytarabine

SUMMARY:
This is a Phase I/II study evaluating safety and efficacy of proteasome inhibitor (bortezomib) in combination with CPX-351 (liposomal daunorubicin and cytarabine) for the treatment of newly-diagnosed TP53-mutated acute myeloid leukemia (TP53m AML).

The primary endpoint of the study is to define safety/tolerability (phase I) and preliminary efficacy profile (phase II) of the treatment. The secondary endpoints of interest are complete remission (CR) rate, detectable minimal residual disease (MRD) status, overall response rate (ORR), rate of allogeneic hematopoietic cell transplantation (allo-HCT), treatment-related mortality (TRM), overall survival (OS), achievement of complete remission anytime in 1 year, and disease-free survival (DFS) at 1 year and 2 years. All the patient outcomes assessments will be performed as part of standard-of-care AML management.

The hypothesis is the combination of bortezomib and CPX-351 will have an acceptable safety profile in this patient population based on the data from previous studies. The treatment will attenuate Nuclear Factor kB pathway activation in these cells and eradicate TP53m leukemia stem cells (LSC) leading to increased response rate and survival in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years at time of consent)
* Have not received any systemic chemotherapy for the treatment of AML. Use of hydroxyurea and leukapheresis to control excess peripheral blasts is permissible. WBC < 25,000 to initiate bortezomib, must reach this threshold by day 7 of CPX-351.
* Karnofsky performance status (KPS) ≥ 70
* Adequate renal, hepatic and cardiac function defined as
* Renal: An estimated glomerular filtration rate ≥ 30 mL/min/1.73 m2
* Hepatic: AST and ALT ≤3 x ULN, ALP ≤2.5 x ULN, and total bilirubin ≤1.5 x ULN. (exception for Gilbert's syndrome or leukemic infiltration of liver)
* Cardiac: New York Heart Association (NYHA) Class I or II, left ventricular ejection fraction > 50% by echocardiogram, MUGA or cardiac MRI
* Sexually active couples of childbearing potential must agree to use effective contraception or abstinence during treatment and for at least 7 months after the final dose of study drug
* Provides voluntary written consent before the performance of any study related activities not part of standard of care.

Exclusion Criteria:

* Received systemic chemotherapy for the treatment of AML
* Bi-phenotypic acute leukemia or mixed lineage leukemia, acute promyelocytic leukemia
* Active central nervous system malignancy or symptoms of CNS involvement
* Symptomatic extramedullary disease
* Known history of uncontrolled HIV or active hepatitis B or active hepatitis C infection
* Has any of the following cardiac abnormalities
* Symptomatic congestive heart failure
* Myocardial infarction less than or equal to 6 months prior to enrollment
* Unstable angina pectoris
* Serious uncontrolled cardiac arrhythmia
* Concomitant malignancies or previous malignancies with less than a 1-year disease free interval at the time of signing consent. Potential participants with adequately resected basal or squamous cell carcinoma of the skin, or adequately resected carcinoma in situ (e.g., cervix) may enroll irrespective of the time of diagnosis
* Participants for whom administration of CPX-351 would exceed their lifetime cumulative daunorubicin exposure limit of 550 mg/m2 (or 400 mg/m2 in patients with prior chest radiation) or equivalent anthracycline dose.
* Pregnant or breastfeeding, or planning pregnancy within 3 months after the treatment completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-01-27 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Complete Response | 2 years
  To evaluate the CR rate of bortezomib + CPX-351 for the treatment of TP53m AML.
Determine Maximum Tolerated Dose | 1 year

SECONDARY OUTCOMES:
Determine Overall Response Rate | 2 years
  Evaluate ORR (CR+CRi) after treatment
Average rate of allo-HCT among participants | 2 years
  Evaluate the rate of allo-HCT within 2 years among patients who received treatment
Overall Survival | 1 year
  estimate 1-year and 2-year OS, defined as the time from cohort assignment to death from any cause
Overall Survival | 2 year
  estimate 1-year and 2-year OS, defined as the time from cohort assignment to death from any cause
Average time to relapse | 2 year
  • To estimate time to relapse, defined as the time from cohort assignment to disease recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States